CLINICAL TRIAL: NCT02521740
Title: Soutien Des Soins Informels Aux Personnes âgées Fragiles : Accompagnement Des Aidants Sur Base d'Une évaluation Clinique et Biologique de la Charge de Soins.
Brief Title: CAREGIVER2, Caregiver's Health Assessment : Clinical and Biological Markers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire UCLouvain Namur (Other)
Collaborators: University of Liege (Other); University of Namur (Other)
Responsible Party: Principal Investigator, Professor Maximilien Gourdin, Directeur Médical adjoint aux missions universitaires, Centre Hospitalier Universitaire UCLouvain Namur
Other Study IDs: 1318184
Record Dates: First submitted 2015-06-29; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Caregivers
Keywords: biological marker; frailty; burden; nutrition; elderly
MeSH Terms: conditions — Frailty | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples taken between 8 and 11 am. Blood parameters including cell counts and assays of acute phase proteins (C-reactive protein (CRP), albumin, pre-albumin) are determined according to the routine of the hospital.
  PBMC are isolated by centrifugation in a Lympho-Ficoll gradient by the biobank of CHU Dinant Godinne.
  Collected plasma is stored at -80 °C until analysis. The amounts of insulin-like growth factor-1 (IGF-1), interleukin-6 (IL-6) are essayed by enzyme-linked immunosorbent assay (ELISA).
  PBMC are sent to Liege (GIGAI3) and Namur (URBC) for respectively ADN and ARN analyses.
  ADN analyses concerned the immunity markers and ARN analyses concerned the transcriptomics and epigenetic markers.
  The biobank of the CHU Dinant-Godinne meets the requirements of the quality book developed by the biobanks of Walonnie-Bruxelles (BWB).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- caregivers: someone who takes care and lives with a disabled elderly
  Interventions: Other: Research questionnaires, blood sample
- controls: someone who lives with an healthy elderly
  Interventions: Other: Research questionnaires, blood sample

INTERVENTIONS:
Other: Research questionnaires, blood sample — assessment of health (frailty, nutrition, physical performance, depression, burden, sense of coherence, caregiver reaction)

SUMMARY:
Providing care for a disabled elderly may represent a risk for the health of the caregiver. The objective of the study is to assess the impact of caregiving in terms of clinical and biological markers in relation to disability and cognitive impairment.

DETAILED DESCRIPTION:
The investigators hypothesize that an accumulation of stressful events related to care giving may induce a stress response to the caregiver. This stress response can be measured by biological markers (inflammation, transcription and immunity) and also by clinical markers (frailty, physical performance, nutrition). This stress response can be influenced by the subjective burden of the caregiver and by the severity of the disease of the care receiver (Activity of daily life capabilities, cognitive function, behavioral disturbance).

ELIGIBILITY:
Inclusion Criteria:

* living with the care-receiver ( or with a healthy elderly for the controls)
* care-receiver dependent for at least one Activity of the daily living ( Katz index) or having cognitive disorder ( >2 Global Deterioration Scale)

Exclusion Criteria:

* institutionalised elderly
* inability to understand and speak french
* Acute disease within the past month
* Anti-inflammatory or immuno-suppressive treatment
* End-of-life care

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: * caregivers of a community dwelling dependent elderly (≥70years)
  * controls : poeple who lives with a healthy elderly (≥70years)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Levels of biomarkers across groups | at baseline
  biomarkers of inflammation (cortisol, high sensitive C-Reactive Protein,Interleukin-6), immunity (TRECS, telomere length) and transcriptomics/epigenetics

SECONDARY OUTCOMES:
Relation between biomarkers, subjective burden and the care receiver situation | at baseline
  biomarkers of inflammation (cortisol, high sensitive C-Reactive Protein,Interleukin-6), immunity (TRECS, telomere length) and transcriptomics/epigenetics and their relations with the Zarit burden, the caregiver reaction assessment, the depression scale and the sense of coherence scale and with the situation of the care receiver ( Katz index, cognitive impairment, behavioral disturbance)

OTHER OUTCOMES:
Relation between biomarkers, subjective burden and the care receiver situation | at baseline
  biomarkers of inflammation (cortisol, high sensitive C-Reactive Protein,Interleukin-6), immunity (TRECS, telomere length) and transcriptomics/epigenetics and their relations with the Zarit burden, the caregiver reaction assessment, the depression scale and the sense of coherence scale and with the situation of the care receiver ( Katz index, cognitive impairment, behavioral disturbance)
comparison of health events | after 12 month
  Institutionalization, increase of formal home help services, hospitalisations
relation between biomarkers at baseline and functional decline | after 12 month
Levels of clinical markers across groups | at baseline and after 12 month
  frailty, physical performance, nutrition, depression
relation between biomarkers at baseline and burden | after 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Marie de Saint-Hubert, MD, PhD, Study Chair — CHUDinant-Godinne
Locations (1):
- CHU Dinant-Godinne, Mont-Godinne, Yvoir, Belgium